CLINICAL TRIAL: NCT06161818
Title: Total Neoadjuvant Therapy for Lymph Node-positive Adenocarcinoma of the OESophagus and Oesophagogastric Junction: a Phase II Study
Brief Title: Total Neoadjuvant Therapy for Lymph Node-positive Adenocarcinoma of the OESophagus and Oesophagogastric Junction
Acronym: TNT-OES-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. B. (Bianca) Mostert, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNT-OES-2; 2025-521158-40-00 (EU CTIS Number)
Record Dates: First submitted 2023-11-09; First posted 2023-12-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Cancer; Adenocarcinoma of the Esophagus
Keywords: Total Neoadjuvant Therapy; Chemotherapy; Chemoradiotherapy
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Intervention Model Description: Arm A: FLOT-CROSS Arm B: CROSS-FLOT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNT FLOT-CROSS (Experimental): Patients allocated to the TNT FLOT-CROSS arm will be treated with 4 cycles of FLOT chemotherapy followed by a response evaluation consisting of a CT-scan and upper endoscopy with bite-on-bite biopsies of the primary tumor site and of any other suspected lesions in the esophagus. Patients with distant metastases will go off-study. All other patients will proceed to CROSS chemoradiotherapy.
  Interventions: Drug: FLOT-CROSS or CROSS-FLOT
- TNT CROSS-FLOT (Experimental): Patients allocated to the TNT CROSS-FLOT arm will be treated with CROSS chemoradiotherapy followed by a response evaluation consisting of a CT-scan and upper endoscopy with bite-on-bite biopsies of the primary tumor site and of any other suspected lesions in the esophagus. Patients with distant metastases will go off-study. All other patients will proceed to FLOT chemotherapy.
  Interventions: Drug: FLOT-CROSS or CROSS-FLOT

INTERVENTIONS:
Drug: FLOT-CROSS or CROSS-FLOT — Randomization between TNT FLOT-CROSS and TNT CROSS-FLOT

SUMMARY:
Both neoadjuvant chemoradiotherapy (CROSS) and neoadjuvant chemotherapy (FLOT) have demonstrated overall survival benefit over surgery alone in esophageal and esophagogastric junction (EGJ) cancer. Despite these survival gains, the prognosis remains poor, especially in patients with nodal-positive adenocarcinoma (cN+ AC) (5-year survival 36%, compared to 55% for cN0). This highlights the need for more effective treatment options, and justifies treatment intensification in these patients.

The aim of this study is to determine the efficacy and feasibility of TNT FLOT-CROSS and TNT CROSS-FLOT in patients with resectable, cN+ AC of the esophagus or EGJ.

DETAILED DESCRIPTION:
This study hypothesizes that the benefits of the locoregional control of CROSS combined with the systemic effect of FLOT leads to better disease control and survival in cN+ AC patients. This Total Neoadjuvant Treatment (TNT) strategy was found to be feasible in the previous TNT-OES-1 trial. The optimal sequence of CROSS and FLOT is yet unknown. Therefore, the hypothesis of this study is that the progression-free survival (PFS) of patients treated with TNT FLOT-CROSS and TNT CROSS-FLOT will be ≥10% compared to the PFS after CROSS in an appropriate historical cohort.

ELIGIBILITY:
Inclusion Criteria:

• Patients with cT2-4aN+M0 resectable adenocarcinoma of the oesophagus or EGJ (Siewert type I-II) according to the 8th edition of the Union for International Cancer Control (UICC) TNM classification for Esophageal Cancer who are planned to undergo nCRT or FLOT (43). In case of stage cT4a, curative resectability has to be explicitly verified by the multidisciplinary tumor board.

Clinical N+ status should be determined by EUS or 18F-FDG PET/CT. Clinical M0 status must be determined by 18F-FDG PET/CT.

* Maximum of 4 cm ingrowth in the cardia, measured by upper endoscopy.
* In case of tumor and/or lymph node involvement below the diaphragm, the most proximal involved lymph node station cannot be higher than N7 (Appendix C).
* In case of no tumor or lymph node involvement below the diaphragm, the most proximal involved lymph node station cannot be higher than N4 (Appendix C).
* Age ≥ 18 years. For patients aged 70 years or older, a geriatric screening tool (G8) should be used to assess functioning across the domains. If a patient has a score of 14 or lower on the G8, a comprehensive geriatric assessment (CGA) should be done prior to inclusion (Appendix D).
* No prior abdominal, thoracic or cervical radiotherapy overlapping with the CROSS irradiation fields.
* No prior cytotoxic chemotherapy for oesophageal cancer.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1 (44).
* Weight loss <10%.
* Adequate cardiac and respiratory function (cardiac or pulmonary function tests such only necessary in symptomatic patients).
* Adequate bone marrow function (White Blood Cells >3x109/L; Haemoglobin >5.5 mmol/L; platelets >100x109/L). In the event of transfusions, the last red blood cell transfusion should be more than 2 weeks before inclusion.
* Adequate renal function (Glomerular Filtration Rate >50 ml/min) or serum creatinine ≤1.5 x upper limit of normal (ULN) and adequate liver function (total bilirubin <1.5x Upper Level of Normal (ULN); Aspartate transaminase (AST) <2.5x ULN and Alanine transaminase (ALT) <3x ULN.
* A negative serum pregnancy test in women of child-bearing potential during screening period.
* Use of adequate contraception during the study up to 3 months after the end of the study.
* Written informed consent and ability to understand the nature of the study and the study-related procedures and to comply with them.

Exclusion Criteria:

* Patients with tumours of squamous, adenosquamous or other non-adenocarcinoma histology.
* Patients who are eligible for and want to participate in the TRAP-2 trial (NCT05188313)
* Patients with overt hematogenous (organ) metastasis, distant lymphatic metastases (cervical/retroperitoneal), peritoneal or pleural dissemination, as detected on 18F-FDG PET/CT or regular CT-scan. In patients in whom a diagnostic laparoscopy is indicated (to assess resectability or to exclude peritoneal disease), tumor-positive cytology peritoneal fluid is also an exclusion criteria.
* Clinically significant (active) cardiac disease (e.g. symptomatic coronary artery disease of myocardial infarction within the last 12 months) or lung disease (forced expiratory volume in one second (FEV1) <1.5L).
* Peripheral neuropathy grade >1, according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (37).
* Homozygous DPYD genotype (tested for *2A, *13, 2846A>T, and 1236G>A)
* Pregnant and lactating women, or patients of reproductive potential who are not using effective contraception. If barrier contraceptives are used, they must be continued by both sexes throughout the study.
* Other active malignancies with a prognosis interfering with that of oesophageal cancer.
* Expected lack of compliance with the protocol.
* Limitations such as language barriers, dementia, or altered mental status that make it impossible for the participant to understand the study, provide informed consent, and complete quality of life questionnaires. Participants who do not speak the primary study language may still be included if the study information is adequately translated or explained (e.g., read aloud in their native language) and they demonstrably understand the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 24 months
  To determine the progression-free survival (PFS) after TNT (both FLOT-CROSS and CROSS-FLOT), the PFS is defined as the time interval from randomization to the first event of locoregional failure after surgery, or locoregional progression leading to irresectability prior to surgery , progression to metastatic disease or death

SECONDARY OUTCOMES:
Feasibility, completion of treatment | 30 months
  To assess the feasibility of TNT FLOT-CROSS and TNT CROSS-FLOT. Feasibility is defined as the proportion of patients that complete all 4 cycles of FLOT and all 5 chemotherapy cycles of CROSS, permitting dose reductions and delays.
Overall survival | 24 months
  To determine the effect of TNT FLOT-CROSS and TNT CROSS-FLOT on overall survival. OS is calculated from the date of randomization to the date of death due to any cause or, for patients alive at trial closure, date of last follow-up
Therapy-related toxicity | 30 months
  The number of patients with any major systemic therapy related toxicity, defined as grade ≥ 3 according to the Common Terminology Criteria for Adverse Events (CTCAE ) version 5.0), up to one month after the last administration of TNT
Dose reductions of TNT | 30 months
  The number of patients requiring dose reductions or treatment delays during CROSS and FLOT
Need of G-CSF | 60 months
  The number of patients requiring G-CSF as primary or secondary prophylaxis
Postoperative morbidity and mortality | 42 months
  To assess the effect of TNT FLOT-CROSS and TNT CROSS-FLOT on postoperative morbidity (Clavien-Dindo ≥3) and 30- and 90-day mortality.
Surgical-related outcomes | 42 months
  To determine the effect of TNT FLOT-CROSS and TNT CROSS-FLOT on surgery-related outcomes (i.e. proportion that proceed to esophagectomy as planned, radical (R0) resection rate).
Non-surgical related outcomes | 30 months
  To determine the effect of TNT FLOT-CROSS and TNT CROSS-FLOT on non-surgical outcomes: the proportion of patients who choose for active surveillance instead of surgery after CRE-2
Clinical response rate | 42 months
  To assess the clinical response rates after TNT FLOT-CROSS and TNT CROSS-FLOT. Clinical complete response (cCR) rate is defined as the percentage of patients without residual locoregional disease or distant metastases at CRE-2, measured by PET-scan and bite-on-bite biopsies with endoscopy and EUS.
Pathological response rate | 42 months
  To assess the pathological response rate after TNT FLOT-CROSS and TNT CROSS-FLOT. Pathological complete response (pCR) rate in those who underwent an oesophagectomy is defined as ypT0N0. Major pathological response in those who underwent oesophagectomy, defined as Mandard 1-2.
Distant metastases | 30 months
  To assess the proportion of distant metastases after TNT FLOT-CROSS and TNT CROSS-FLOT at 6 weeks after completion of treatment
Quality of life assessed by EORTC-C30 | 42 months
  The quality of life will be assessed with the EORTC-C30 questionnaire
Quality of life assessed by EORTC QLQ-OG25 | 42 months
  To determine the effect of TNT FLOT-CROSS and TNT CROSS-FLOT on quality of life, assessed by the QoL questionnaires: EORTC QLQ-OG25
The PD-L1 combined positive score (CPS) | 42 months
  The PD-L1 combined positive score (CPS) of TNT FLOT-CROSS and TNT CROSS-FLOT before treatment and in metastases. The PD-L1 CPS will be measured as a continuous variable. This will be measured using the 28-8 monoclonal antibody.
Predictive biomarkers | 63 months
  To collect blood at baseline, first clinical response evaluation (CRE-1), CRE-2 and postoperatively to enable future ctDNA based translational studies looking for biomarkers predictive of disease recurrence and early response.
Future ctDNA analysis | 63 months
  To collect tissue at baseline, CRE-1, CRE-2 and resection to enable future ctDNA based translational studies looking for biomarkers predictive of disease recurrence and early response.

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Mostert, MD, PhD, Principal Investigator — Erasmus Medical Centre
Locations (10):
- Netherlands (10):
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Frisius medisch centrum, Leeuwarden, North Brabant
  - Elisabeth Tweesteden Ziekenhuis, Tilburg, North Brabant
  - Amsterdam UMC, Amsterdam, North Holland
  - Erasmus Medical Centre, Rotterdam, South Holland
  - Ziekenhuisgroep Twente, Almelo
  - Antoni van Leeuwenhoek/Nederlands Kanker Instituut, Amsterdam
  - Gelre ziekenhuis, Apeldoorn
  - Leids Universitair Medisch Centrum, Leiden
  - Radboud Universitair Medisch Centrum, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Zijden CJ, Eyck BM, van der Gaast A, van Doorn L, Nuyttens JJME, van Lanschot JJB, Wijnhoven BPL, Mostert B, Lagarde SM. Chemotherapy aNd chemoradiotherapy for adenocarcinoma of the OESophagus and esophagogastric junction with oligometastases: Protocol of the TNT-OES-1 trial. Contemp Clin Trials Commun. 2022 May 28;28:100934. doi: 10.1016/j.conctc.2022.100934. eCollection 2022 Aug. PMID 35669486